CLINICAL TRIAL: NCT01328743
Title: Brief Alcohol Intervention for HIV-Infected Men Who Have Sex With Men (MSM) in a Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Peter Monti, Professor of Behavioral and Social Sciences, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIAAA-P01-AA019072-1
Record Dates: First submitted 2011-03-31; First posted 2011-04-05 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Hazardous Drinking; HIV
MeSH Terms: interventions — Ethanol; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as usual (No Intervention): Treatment as usual in an HIV primary care setting. Participants receive assessment of alcohol use but not counseling or advice regarding drinking.
- Brief Alcohol Intervention (Experimental): Participants receive 3 face-to-face sessions of counseling on alcohol use and 2 follow-up phone calls
  Interventions: Behavioral: Brief alcohol intervention

INTERVENTIONS:
Behavioral: Brief alcohol intervention — 3 sessions of individual face-to-face counseling at baseline, 3 and 6 months. Sessions are motivationally focused including discussion of pros and cons of drinking and feedback on health and its relation to heavy drinking
  Arms: Brief Alcohol Intervention

SUMMARY:
This is a randomized clinical trial to examine the effects of a brief counseling intervention for heavy drinking HIV-infected men who have sex with men compared to HIV care as usual. The study tests the hypothesis that brief counseling will lower drinking in these patients and that reductions in drinking will be associated with better HIV-related outcomes.

DETAILED DESCRIPTION:
This study is a randomized clinical trial in which 224 heavy drinking men who have sex with men (MSM), who receive their HIV primary care at Fenway Health in Boston, are randomly assigned to treatment as usual (TAU) or TAU plus a brief intervention to reduce alcohol use (TAU-BI). TAU-BI will be based in Motivational Interviewing and include personalized feedback tailored to an HIV-infected MSM population. Follow-ups will occur at 3, 6, and 12 months. The first primary aim of the study is to test the hypothesis that TAU-BI, compared to TAU, will result in reduced alcohol consumption over a 12-month follow-up period as indicated by: (1) a lower number of alcoholic drinks consumed per week; (2) a lower number of drinking days within each follow-up period; and (3) a lower number of heavy drinking days within each follow-up period. The second primary aim is to test the hypothesis that greater reductions in alcohol use will be associated with (1) greater adherence to HIV medication regimens; (2) less engagement in high-risk sexual behavior that could result in HIV transmission; (3) lower plasma HIV RNA levels (viral load) (CD4 cell counts will be a secondary outcome in this sub-aim); (4) improved liver function tests; and (5) improved neurocognitive function.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* drink heavily at least once per month on average (≥5 drinks) or drink more than 14 drinks per week
* have a confirmed diagnosis of HIV/AIDS
* be a male who has had sex (oral or anal) with a male partner in the past 3 months.

Exclusion Criteria:

* current intravenous drug use
* currently psychotic, suicidal, or manic
* are currently being treated or have been treated in the past 3 months for an HIV-related opportunistic infection
* currently receiving treatment for an alcohol or drug problem

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-05; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Monti, Ph.D., Principal Investigator — Brown University; Christopher Kahler, Ph.D., Study Director — Brown University
Locations (1):
- Fenway Health, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Zelaya DG, Guy AA, Surace A, Mastroleo NR, Pantalone DW, Monti PM, Mayer KH, Kahler CW. Modeling the Impact of Race, Socioeconomic Status, Discrimination and Cognitive Appraisal on Mental Health Concerns Among Heavy Drinking HIV+ Cisgender MSM. AIDS Behav. 2022 Dec;26(12):3925-3938. doi: 10.1007/s10461-022-03719-0. Epub 2022 Jun 10. PMID 35687187

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment as Usual | Brief Alcohol Intervention
Started | 91 | 89
Completed | 82 | 79
Not Completed | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | Brief Alcohol Intervention | Total
Number analyzed (Participants) | 91 | 89 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (10.5) | 41.0 (10.3) | 42.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 91 | 89 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 31
  Not Hispanic or Latino | 76 | 73 | 149
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 14 | 35
  White | 64 | 70 | 134
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 91 | 89 | 180

OUTCOME MEASURES:

1. Primary Outcome: Number of Alcoholic Drinks Consumed
Description: Number of standard alcoholic drinks consumed per week in the past month
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: drinks per week
Arm/Group | Treatment as Usual | Brief Alcohol Intervention
Number analyzed (Participants) | 82 | 79
drinks per week | 11.6 [4.2 to 21.5] | 7.2 [2.3 to 12.6]
Statistical Analysis 1: Comparison: Treatment as Usual; Test type: Superiority; p = .04, t-test, 2 sided

2. Primary Outcome: Number of Heavy Drinking Days
Description: Number of heavy drinking days (drinking 5 or more drinks in a day) in the past month
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Treatment as Usual | Brief Alcohol Intervention
Number analyzed (Participants) | 82 | 79
Days | 3 [1 to 6] | 1 [0 to 3]
Statistical Analysis 1: Comparison: Treatment as Usual; Test type: Superiority; p < .01, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Number of Heavy Drinking Days
Description: Number of heavy drinking days (drinking 5 or more drinks in a day) in the past month
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Treatment as Usual | Brief Alcohol Intervention
Number analyzed (Participants) | 86 | 78
Days | 4 [1 to 9] | 2 [0 to 4]
Statistical Analysis 1: Comparison: Treatment as Usual; Test type: Superiority; p < .01, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Number of Heavy Drinking Days
Description: Number of heavy drinking days (drinking 5 or more drinks in a day) in the past month
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Treatment as Usual | Brief Alcohol Intervention
Number analyzed (Participants) | 88 | 79
Days | 4 [1 to 9] | 3 [1 to 8]
Statistical Analysis 1: Comparison: Treatment as Usual; Test type: Superiority; p = .48, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Number of Alcoholic Drinks Consumed
Description: Number of standard alcoholic drinks consumed per week in the past month
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: drinks per week
Arm/Group | Treatment as Usual | Brief Alcohol Intervention
Number analyzed (Participants) | 88 | 79
drinks per week | 14.4 [7.6 to 27.3] | 11.9 [6.5 to 19.6]
Statistical Analysis 1: Comparison: Treatment as Usual; Test type: Superiority; p = .25, t-test, 2 sided

6. Primary Outcome: Number of Alcoholic Drinks Consumed
Description: Number of standard alcoholic drinks consumed per week in the past month
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: drinks per week
Arm/Group | Treatment as Usual | Brief Alcohol Intervention
Number analyzed (Participants) | 86 | 78
drinks per week | 14.5 [4.7 to 26.4] | 8.0 [4.2 to 12.8]
Statistical Analysis 1: Comparison: Treatment as Usual; Test type: Superiority; p < .001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Treatment as Usual | Brief Alcohol Intervention
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/89
Other Adverse Events (participants affected / at risk) | 0/91 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes